CLINICAL TRIAL: NCT00529841
Title: A Novel Therapeutic Modality for Congenital Adrenal Hyperplasia
Brief Title: Research Study for Children With Salt Wasting Congenital Adrenal Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-19704; GCRC # 0962 (Other: Baylor College of Medicine)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Adrenal Hyperplasia, Congenital
Keywords: Salt Wasting Congenital Adrenal Hyperplasia; Subcutaneous Hydrocortisone
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — hydrocortisone hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Hydrocortisone sodium acetate) (Experimental): Subcutaneous administration of Hydrocortisone sodium acetate via insulin pump
  Interventions: Drug: Hydrocortisone sodium acetate

INTERVENTIONS:
Drug: Hydrocortisone sodium acetate — Subcutaneous administration of medication via insulin pump
  Other Names: Solu-Cortef injection

SUMMARY:
The purpose of this study is to develop a more physiological approach to the management of children and adolescents with salt wasting Congenital Adrenal Hyperplasia.

We will administer the glucocorticosteroid via insulin infusion pump to see whether this treatment will improve the serum hormone concentrations.

DETAILED DESCRIPTION:
The adrenal gland is a small organ of the body. It produces very important chemicals called hormones. One of these hormones, cortisol (the stress hormone) helps the body fight diseases. The other hormone is the aldosterone helps to maintain the normal amount of salt and water in the body. The third type of hormones are the androgens or male hormones, which cause some of the changes during puberty, like the growth of body hair and pimples.

The salt wasting Congenital Adrenal Hyperplasia or CAH disease is a disease of the adrenal gland. Patients with this disease cannot make cortisol or the aldosterone. As a result, their body cannot fight diseases and cannot keep normal amounts of salt and water in the body. At the same time, the gland makes too much of the male hormones, which is bad for the body because too much male hormone slows down growth, increases the growth of body hair, and causes pimples and abnormal period in girls.

Patients with this disease have to take medications every day. However, the treatment does not work very well, because usually the patients do not have the right amount of hormone in their body. Usually the body gets too much hormone right after taking the pills. A couple of hours later the body has too little of the hormones, because in the meantime the body gets rid of the medication.The healthy adrenal gland makes the hormones throughout the day in different amounts. The patients with this disease take the medication only a couple of times a day. They take the Florinef tablet once a day and the Cortisol tablet two or three times a day. The treatment that we use today by mouth cannot copy the natural hormone productions of the adrenal gland. Because of this it does not make much of a difference in the patient's life.

We would like to improve the treatment and find out the effect of a new treatment. In this study we will try to imitate the body's normal hormone production and will give the medication via an insulin pump to see if this treatment method will decrease the male hormones in the blood. This study will help us to develop a new and better treatment for children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Children with salt wasting CAH otherwise healthy without other chronic disease
* Age: between 3 and 18 years of age
* Body weight 23 kg (50 lbs) or above
* Hemoglobin equal to or higher than 12 g/dl before the study
* Supportive family environment

Exclusion Criteria:

* Age less than 3 or older than 18 years at the time of study
* Other chronic disease
* Hemoglobin less than 12 g/dl
* Non-supportive family
* Allergy to local anesthetics

Criteria for study termination: If the subject's parents are unable to manage/operate the pump, the subject will be withdrawn from the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Serum 17-OHP concentration in the morning | 11 days

SECONDARY OUTCOMES:
serum steroid hormone profiles | 11 days
serum blood glucose | study days 2,3 and 11
serum sodium | study days 2,3 and 11

CONTACTS AND LOCATIONS:
Overall Officials: Morey W Haymond, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- BCM, Texas Children's Hospital Clinic and General Clinical Research Center, Houston, Texas, United States

REFERENCES:
- [Background] Esteban NV, Loughlin T, Yergey AL, Zawadzki JK, Booth JD, Winterer JC, Loriaux DL. Daily cortisol production rate in man determined by stable isotope dilution/mass spectrometry. J Clin Endocrinol Metab. 1991 Jan;72(1):39-45. doi: 10.1210/jcem-72-1-39. PMID 1986026
- [Background] Kerrigan JR, Veldhuis JD, Leyo SA, Iranmanesh A, Rogol AD. Estimation of daily cortisol production and clearance rates in normal pubertal males by deconvolution analysis. J Clin Endocrinol Metab. 1993 Jun;76(6):1505-10. doi: 10.1210/jcem.76.6.8501158.
- [Background] Speiser PW. Toward better treatment of congenital adrenal hyperplasia. Clin Endocrinol (Oxf). 1999 Sep;51(3):273-4. doi: 10.1046/j.1365-2265.1999.00780.x. No abstract available. PMID 10469004
- [Background] Cutler GB Jr, Laue L. Congenital adrenal hyperplasia due to 21-hydroxylase deficiency. N Engl J Med. 1990 Dec 27;323(26):1806-13. doi: 10.1056/NEJM199012273232605. No abstract available. PMID 2247119
- [Background] Winterer J, Chrousos GP, Loriaux DL, Cutler GB Jr. Effect of hydrocortisone dose schedule on adrenal steroid secretion in congenital adrenal hyperplasia. J Pediatr. 1985 Jan;106(1):137-42. doi: 10.1016/s0022-3476(85)80486-8. PMID 3871229
- [Background] Wallace WH, Crowne EC, Shalet SM, Moore C, Gibson S, Littley MD, White A. Episodic ACTH and cortisol secretion in normal children. Clin Endocrinol (Oxf). 1991 Mar;34(3):215-21. doi: 10.1111/j.1365-2265.1991.tb00297.x. PMID 1645237
- [Background] Merza Z, Rostami-Hodjegan A, Memmott A, Doane A, Ibbotson V, Newell-Price J, Tucker GT, Ross RJ. Circadian hydrocortisone infusions in patients with adrenal insufficiency and congenital adrenal hyperplasia. Clin Endocrinol (Oxf). 2006 Jul;65(1):45-50. doi: 10.1111/j.1365-2265.2006.02544.x. PMID 16817818
- [Background] Lukert BP. Editorial: glucocorticoid replacement--how much is enough? J Clin Endocrinol Metab. 2006 Mar;91(3):793-4. doi: 10.1210/jc.2005-2737. No abstract available. PMID 16522704
- [Background] Claude J.Migeon. Can the Long Range Results of the Treatment of Congenital Adrenal Hyperplasia be improved? JCEM 1996 Vol 81, No 9 3187-3189
- [Background] Laue L, Merke DP, Jones JV, Barnes KM, Hill S, Cutler GB Jr. A preliminary study of flutamide, testolactone, and reduced hydrocortisone dose in the treatment of congenital adrenal hyperplasia. J Clin Endocrinol Metab. 1996 Oct;81(10):3535-9. doi: 10.1210/jcem.81.10.8855797.
- [Background] Mah PM, Jenkins RC, Rostami-Hodjegan A, Newell-Price J, Doane A, Ibbotson V, Tucker GT, Ross RJ. Weight-related dosing, timing and monitoring hydrocortisone replacement therapy in patients with adrenal insufficiency. Clin Endocrinol (Oxf). 2004 Sep;61(3):367-75. doi: 10.1111/j.1365-2265.2004.02106.x. PMID 15355454
- [Background] Sheila K.Gunn et al Subcutaneous Hydrocortisone Delivery mimics Physiologic Cortisol Concentrations, Poster, Endocrine Society Meeting 2000